CLINICAL TRIAL: NCT00968331
Title: Study of Lenalidomide(Revlimid) Plus Rituximab (Revlirit Regimen) in Elderly Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The EC withdrawn the approval becuase of possible conflicts of interests between our Institute and Supporter (Celgene)
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Pier Luigi Zinzani, Professor, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REVLIRIT01
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: relapsed and refractory DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Lenalidomide; Rituximab

ARMS (1):
- REVLIMID plus RITUXIMAB (Experimental): Oral Lenalidomide is initiated on day 1 of cycle 1 at the dose of 20 mg daily for 21 days with 7 days rest (28 day cycle) for a total of 4 cycles.
  Rituximab is administered on day 1 and day 21 of each cycle at the dose of 375 mg/m2 for a total of 4 cycles.
  Interventions: Drug: Lenalidomide plus Rituximab

INTERVENTIONS:
Drug: Lenalidomide plus Rituximab — Oral Lenalidomide is initiated on day 1 of cycle 1 at the dose of 20 mg daily for 21 days with 7 days rest (28 day cycle) for a total of 4 cycles. Rituximab is administered on day 1 and day 21 of each cycle at the dose of 375 mg/m2 for a total of 4 cycles.

SUMMARY:
Oral Lenalidomide is initiated on day 1 of cycle 1 at the dose of 20 mg daily for 21 days with 7 days rest (28 day cycle) for a total of 4 cycles. Rituximab is administered on day 1 and day 21 of each cycle at the dose of 375 mg/m2 for a total of 4 cycles.

After this induction phase, the CR, PR and SD will continue Lenalidomide with the same schedule for other 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Be = 65 years of age at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Patients with histological confirmation of DLBCL.
* Stage of disease at study entry may include stage II-III-IV according to Ann Arbor Classification
* Patients must have failed at least one prior treatments
* ECOG performance status of equal or less than 2 at study entry
* nLaboratory test results within these ranges:
* Absolute neutrophil count equal or major than 1.0 x 109/L
* Platelet count equal or major than 50 x 109/L
* Serum creatinine equal or less than 2.0 mg/dL
* Total bilirubin equal or less than 1.5 mg/dL
* AST (SGOT) and ALT (SGPT) equal or less than 2 x ULN or equal or less 5 x ULN if hepatic metastases are present
* Hemoglobin equal or major than 8 g/dl
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study:

  1. for at least 28days before starting study drug
  2. while participating in the study
  3. for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom,diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Disease free of prior malignancies for equal or major 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the antitumour activity of Lenalidomide plus Rituximab (REVLIRIT) as salvage treatment in elderly patients with relapsed or refractory DLBCL, in terms of Overall Response Rate (CR and PR) | 12 months

SECONDARY OUTCOMES:
To assess the overall feasibility of the REVLIRIT regimen in terms of response To assess the duration of response, TTP and PFS, safety and tolerability of the REVLIRIT regimen in terms of AE and SAE frequency and severity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Of Hematology "Seràgnoli", Bologna, Italy